CLINICAL TRIAL: NCT01209806
Title: The Effects of Moviprep With Simethicone on Colonic Bubbles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: #09D.472
Record Dates: First submitted 2010-07-12; First posted 2010-09-27 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Bubbles in Colon at Time of Colonoscopy
MeSH Terms: interventions — Simethicone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- simethicone (Active Comparator)
  Interventions: Drug: simethicone
- no simethicone (No Intervention)

INTERVENTIONS:
Drug: simethicone — 400 mg simethicone at 6pm night prior to colonoscopy 400 mg simethicone 4 hours before colonoscopy
  Other Names: Alka-Seltzer® Gas Relief Maximum Strength Softgels®; Flatulex® Drops; GasAid® Maximum Strength Softgels®; Gas-X®; Gas-X® Extra Strength; Gas-X® Extra Strength Liquid; Gas-X® Extra Strength Softgels®; Genasyme®; Genasyme® Drops; Maalox® Anti-Gas Extra Strength; Maalox® Anti-Gas Regular Strength; Mylanta® Gas Relief; Mylanta® Gas Relief Gelcaps®; Mylanta® Gas Relief Maximum Strength; Mylicon® Infant's Drops; Phazyme® Infant Drops; Phazyme®-125 Softgels®; Phazyme®-166 Maximum Strength; Phazyme®-166 Maximum Strength Softgels®
  Arms: simethicone

SUMMARY:
The purpose of this study is to determine whether the administration of PEG along with simethicone will reduce the incidence of colonic bubbles that interfere with polyp detection.

DETAILED DESCRIPTION:
evaluating if simethicone is better than placebo at decreasing gas in the colon at time of colonoscopy so that it is easier for the endoscopist to see polyps

ELIGIBILITY:
Inclusion Criteria:

-Elective outpatients undergoing colonoscopy using split dose PEG-ELS with sodium ascorbate and ascorbic acid

Exclusion Criteria:

* Unable or unwilling to give informed consent
* Age < 18 years
* Pregnant
* Breast feeding
* Established or suspected gastroparesis
* Pseudo-obstruction - established or suspected
* Severe constipation (< 1 BM a week)
* Bowel obstruction
* Greater than 50% resection of colon
* Chronic nausea or vomiting
* Consumed > 100% standard dose of PEG-ELS (i.e. more than 2L)
* G6PD deficiency
* PEG allergy
* Significant psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Efficacy - Entire colon | At time of colonoscopy
  Successful cleansing defined as score or excellent or good Unsuccessful cleansing defined as score of fair or inadequate

SECONDARY OUTCOMES:
Efficacy - Right colon | At time of colonoscopy
  Successful cleansing defined as score or excellent or good Unsuccessful cleansing defined as score of fair or inadequate
Adenoma detection | at time of colonoscopy
  Defined as number of adenoma/patient Secondarily evaluate % of patients with at least 1 adenoma
Flushing | at time of colonoscopy
  Defined as need for any (1, 2, or 3) flushing
  • 0 = none, 1 = <50 ml, 2 = 50-100 ml, 3 = >100 ml
Tolerance | during prep ingestion
  Prep completion
  • Completion defined as consuming > 90%
  Sleep
  * Primary definition as quality of sleep
  * Also evaluate duration of sleep Overall satisfaction
  * Use visual analogue (Likert) scale Adverse events - nausea, vomiting, abdominal pain, bloating, light-headedness
  * Primary is incidence
  * Secondary is severity using Likert scale
Safety | at time of colonoscopy
  Vitals with orthostatic measures (BP, Pulse) day of colonoscopy Physical exam

CONTACTS AND LOCATIONS:
Overall Officials: David Kastenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States